CLINICAL TRIAL: NCT03048409
Title: Retrospective Tube Feeding Tolerance in Adults With Intolerance After Switch to a Peptide-based Formula
Acronym: RAP
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 16.06.US.HCN
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Enteral Feeding Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enteral tube fed adults: Enteral formula
  Interventions: Other: Enteral Formula

INTERVENTIONS:
Other: Enteral Formula — Enteral feeding with a peptide-based formula.

SUMMARY:
A retrospective chart review to assess feeding tolerance in adults who had been switched from an intact protein formula to a peptide-based formula due to feeding intolerance in a complex continuing care facility.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age on admission to facility
* Prescribed enteral nutrition with the goal to provide at least 90% of estimated daily calorie and protein requirements for ≥ 2 weeks prior to switch
* Received enteral nutrition with an intact protein formula for a minimum of three days prior to a switch to a peptide-based formula
* Have documentation of intolerance to an intact protein formula, followed by a switch in formula received to a peptide-based formula
* Receiving a peptide-based formula formula for ≥ 2 weeks
* Have documentation of an assessment of feeding tolerance following the switch
* Formulas received must be indicated for use in adults.

Exclusion Criteria:

* Abdominal surgery (within past 30 days prior to switch)
* Having any infection, including upper respiratory, viral, gastroenteritis,wound infections, c difficile, at time of switch
* Having documented cow's milk protein allergy at time of switch
* Medical records lacking information on rationale for switch to a peptide-based formula and/or response to change (positive, neutral or negative).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population studied retrospectively will be adult patients in a chronic care facility dependent on enteral nutrition for 90% or more of their nutritional needs and meeting the inclusion/ exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Feeding tolerance - Gastric residuals | Up to 30 days after formula switch
  no change, tolerance improved, tolerance worsened
Feeding tolerance - gagging/retching | Up to 30 days after formula switch
  no change, tolerance improved, tolerance worsened
Feeding tolerance - abdominal distension/gas | Up to 30 days after formula switch
  no change, tolerance improved, tolerance worsened
Feeding tolerance - vomiting | Up to 30 days after formula switch
  no change, tolerance improved, tolerance worsened
Feeding tolerance - stool consistency issues | Up to 30 days after formula switch
  too hard, too loose
Volume of formula consumed in a day vs. goal | Up to 30 days after formula switch
  documentation of feeding volume after switch as "less than," "about the same as," or "more than" feeding volume achieved before switch
Tube feeding interruptions | Up to 30 days after formula switch
  Number of tube feeding interruptions

SECONDARY OUTCOMES:
Weight | Prior to and up to 30 days following formula switch.
  Measured body weight
Medication use | Prior to and up to 30 days following formula switch.
  Documented medication use
Caloric intake | Up to 30 days after formula switch
  Measured daily calorie intake
Protein intake | Up to 30 days after formula switch
  Measured daily protein intake

CONTACTS AND LOCATIONS:
Overall Officials: Jean Chouinard, MD, Principal Investigator — St Vincent's Hospital
Locations (1):
- Bruyere Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No